CLINICAL TRIAL: NCT02917642
Title: Clinical Evaluation of the Effect of Passive Ultrasonic Irrigation on the Reduction of Bacteria and Endotoxins in Root Canals
Brief Title: Effect of Passive Ultrasonic Irrigation on the Reduction of Bacteria and Endotoxins in Root Canals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ericka Tavares Pinheiro, PhD, University of Sao Paulo
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: FAPESP2013/02923-9
Record Dates: First submitted 2016-09-15; First posted 2016-09-28 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Tooth, Nonvital
Keywords: bacterial infection; endotoxin; passive ultrasonic irrigation; root canal treatment
MeSH Terms: conditions — Tooth, Nonvital; Bacterial Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Passive Ultrasonic Irrigation Protocol (Experimental): ultrasonic activation of antimicrobial solutions
  Interventions: Device: Ultrasonic Irrigation
- Non-Ultrasonic Irrigation Protocol (Active Comparator): no-activation of antimicrobial solutions
  Interventions: Device: Non-Ultrasonic Irrigation

INTERVENTIONS:
Device: Ultrasonic Irrigation — Passive Ultrasonic Irrigation is based on the transmission of acoustic energy through the irrigant by a stainless steel wire or endodontic file
  Arms: Passive Ultrasonic Irrigation Protocol
Device: Non-Ultrasonic Irrigation — Syringe and needle irrigation with no-ultrasonic activation
  Arms: Non-Ultrasonic Irrigation Protocol

SUMMARY:
The purpose of this clinical study was to compare the effectiveness of passive ultrasonic irrigation with that of traditional syringe irrigation on the removal of bacteria and endotoxin (lipopolysaccharide [LPS]) from root canals.

DETAILED DESCRIPTION:
Forty teeth with apical periodontitis were randomly allocated into two groups according to the irrigation protocol, passive ultrasonic irrigation (PUI, n = 20) and syringe and needle irrigation (NI, n = 20). Microbiological sampling was performed before (S1) and after the root canal preparation (S2), after the tested irrigation protocols (S3). Total bacteria counts were determined by a quantitative PCR (qPCR) assay; and the endotoxin levels by the LAL assay.

ELIGIBILITY:
Inclusion Criteria:

* Teeth with necrotic pulps and asymptomatic apical periodontitis

Exclusion Criteria:

* patients who had received antibiotics during the previous 3 months or had any general disease,
* teeth that could not be properly isolated with rubber dam,
* non-restored teeth,
* periodontal pockets depths greater than 4 mm,
* previous endodontic treatment,
* open apex,
* crown/root fracture
* root resorption or calcifications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-01; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Gavini, DDS, Ms, PhD, Study Chair — Department of Dentistry, School of Dentistry, University of São Paulo.

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who had received endodontic intervention or declined to participate before assignment: 16 out of 66 patients were excluded from this study.
Period: Overall Study
Arm/Group | Passive Ultrasonic Irrigation Protocol | Non-Ultrasonic Irrigation Protocol
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: teeth
Groups:
- Total: Total of all reporting groups
Arm/Group | Passive Ultrasonic Irrigation Protocol | Non-Ultrasonic Irrigation Protocol | Total
Number analyzed (Participants) | 25 | 25 | 50
Number analyzed (teeth) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 38 [18 to 63] | 34 [18 to 58] | 34 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 8 | 5 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Levels
Description: Quantitative data of total bacterial counts determined by a DNA-based qPCR (quantitative polymerase chain reaction) assay
Time Frame: Through study completion, an average of 2 years
Measure: Median (Full Range); unit: DNA copies
Arm/Group | Passive Ultrasonic Irrigation Protocol | Non-Ultrasonic Irrigation Protocol
Number analyzed (Participants) | 25 | 25
DNA copies | 4290 [0 to 22200] | 10800 [0 to 338000]
Statistical Analysis 1: Comparison: Passive Ultrasonic Irrigation Protocol vs Non-Ultrasonic Irrigation Protocol; The null hypothesis is that the irrigation protocol used after the chemo-mechanical preparation does not influence the reduction of bacteria within the root canal system; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Endotoxin Levels
Description: Quantitative data of endotoxin levels determined by the quantitative kinetic turbidimetric LAL assay
Time Frame: Through study completion, an average of 2 years
Measure: Median (Full Range); unit: EU/mL
Arm/Group | Passive Ultrasonic Irrigation Protocol | Non-Ultrasonic Irrigation Protocol
Number analyzed (Participants) | 22 | 23
EU/mL | 6.53 [0 to 19.4] | 5.75 [0 to 14.8]
Statistical Analysis 1: Comparison: Passive Ultrasonic Irrigation Protocol vs Non-Ultrasonic Irrigation Protocol; The null hypothesis is that the irrigation protocol used after the chemo-mechanical preparation does not influence the reduction of endotoxin within the root canal system; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed because the endodontic treatment does not cause mortality or serious adverse events.
Arm/Group | Passive Ultrasonic Irrigation Protocol | Non-Ultrasonic Irrigation Protocol
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT02917642/Prot_SAP_000.pdf